CLINICAL TRIAL: NCT07338877
Title: RenewDisc Trial: A Prospective Observational Study Comparing Endoscopic Discectomy and Autologous Mesenchymal Stem Cell Therapy in Patients With Discogenic Low Back Pain
Brief Title: RenewDisc Trial: Endoscopic Discectomy and Autologous Stem Cell Therapy for Discogenic Low Back Pain
Acronym: RENEWDISC
Status: Enrolling by invitation | Type: Observational
Sponsor: Europainclinics z.ú. (Other)
Collaborators: Slovak Academy of Sciences (Other Government); Pavol Jozef Safarik University (Other)
Responsible Party: Sponsor
Other Study IDs: 10148/2024/ODDZ-44592
Record Dates: First submitted 2026-01-04; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Discogenic Low Back Pain; Intervertebral Disc Degeneration; Lumbar Disc Disease; Chronic Low Back Pain
Keywords: Discogenic Low Back Pain; Endoscopic Discectomy; Mesenchymal Stem Cells; Regenerative Spine Therapy; Lumbar Intervertebral Disc; Minimally Invasive Spine Surgery
MeSH Terms: conditions — Intervertebral Disc Degeneration; Intervertebral disc disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Endoscopic Discectomy Plus Mesenchymal Stem Cell Therapy: Patients with clinically confirmed discogenic low back pain who undergo transforaminal endoscopic discectomy combined with autologous mesenchymal stem cell application as part of routine clinical care. Treatment selection is based on standard clinical decision-making and is not assigned by the study protocol.
- Endoscopic Discectomy: Patients with clinically confirmed discogenic low back pain who undergo transforaminal endoscopic discectomy as part of standard clinical practice. The study prospectively observes clinical, functional, and imaging outcomes without assigning treatment.
- Endoscopic Mesenchymal Stem Cell Therapy: Patients with clinically confirmed discogenic low back pain who undergo standalone endoscopic application of autologous mesenchymal stem cells as part of routine clinical care. Outcomes are observed prospectively without protocol-driven treatment allocation.

SUMMARY:
he RenewDisc Trial is a prospective observational clinical study evaluating outcomes in patients with confirmed discogenic low back pain who undergo standard clinical care using endoscopic spine procedures. The study observes and compares clinical, functional, and imaging outcomes following endoscopic discectomy, endoscopic discectomy combined with autologous mesenchymal stem cell therapy, or standalone endoscopic application of autologous mesenchymal stem cells.

Participants are treated according to routine clinical decision-making, and no interventions are assigned by the study protocol. Data are collected prospectively at predefined follow-up intervals to assess pain intensity, functional disability, quality of life, and structural changes on magnetic resonance imaging.

DETAILED DESCRIPTION:
Discogenic low back pain is a frequent cause of chronic disability and remains challenging to treat when conservative management fails. Endoscopic spine techniques have emerged as minimally invasive options that allow targeted treatment of disc pathology with reduced tissue trauma. In parallel, regenerative approaches using autologous mesenchymal stem cells have gained interest due to their potential biological effects on disc degeneration.

The RenewDisc Trial is designed as a prospective observational cohort study to systematically collect and analyze real-world clinical data from patients with confirmed discogenic low back pain who undergo endoscopic spine procedures as part of routine clinical care. The study does not assign or randomize treatments. All therapeutic decisions, including the choice of procedure, are made independently by the treating physician based on standard clinical indications and patient preference.

Patients included in the study undergo one of the following standard clinical approaches: endoscopic discectomy, endoscopic discectomy combined with autologous mesenchymal stem cell application, or standalone endoscopic application of autologous mesenchymal stem cells. These approaches represent established clinical practices at participating centers. The study observes outcomes associated with each approach without altering standard care pathways.

Clinical outcomes are assessed prospectively using validated patient-reported outcome measures, including pain intensity scales, functional disability, and health-related quality of life. Imaging follow-up with magnetic resonance imaging is performed at predefined intervals to evaluate structural changes of the intervertebral disc. In patients undergoing bone marrow aspiration as part of standard care, cellular characteristics of the aspirate are analyzed descriptively.

Data are collected at baseline and during scheduled follow-up visits and are recorded using anonymized, randomly generated participant identifiers. The study aims to provide comparative real-world evidence on clinical, functional, and imaging outcomes associated with contemporary endoscopic and regenerative spine treatment strategies for discogenic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Clinical diagnosis of discogenic low back pain
* Positive provocative discography of the target intervertebral disc
* Negative medial branch block
* Preserved lumbar intervertebral disc height greater than 50%
* Pfirrmann grade I-II on lumbar spine MRI
* Back pain with or without radicular pain
* Back pain representing at least 30% of the patient's total reported pain

Exclusion Criteria:

* Lumbar intervertebral disc height reduction greater than 50%
* Presence of Schmorl's nodes in adjacent vertebrae
* Acute or chronic infection
* Presence of hematological disorders
* Back pain representing less than 30% of the patient's total reported pain
* Contraindication to endoscopic spine procedures
* Refusal or inability to provide written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of adult patients with clinically confirmed discogenic low back pain who are evaluated and treated in specialized spine and pain management centers. Eligible participants have imaging and diagnostic findings consistent with early-stage lumbar intervertebral disc degeneration and are considered suitable candidates for endoscopic spine procedures as part of routine clinical care. Patients are enrolled consecutively based on predefined inclusion and exclusion criteria, without protocol-driven treatment assignment.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index (ODI) | From baseline to 24 months after the procedure
  Outcome Measure Description:
  The ODI is a validated 10-item, self-administered questionnaire assessing back-specific functional disability. Total score is converted to a 0-100 scale; higher scores indicate greater disability.
Change From Baseline in Numerical Rating Scale (NRS) for Back Pain | From baseline to 24 months after the procedure
  The Numerical Rating Scale (NRS) is a patient-reported measure of pain intensity ranging from 0 (no pain) to 10 (worst imaginable pain). Patients rate their average back pain intensity at each assessment time point.
Change From Baseline in Visual Analog Scale (VAS) for Leg Pain | From baseline to 24 months after the procedure
  The Visual Analog Scale (VAS) is a 10-cm continuous scale used to assess pain intensity, anchored by "no pain" (0) and "worst imaginable pain" (10).
Magnetic Resonance Imaging (MRI) Assessment of Intervertebral Disc Morphology | At 6, 12, and 24 months after the procedure
  MRI evaluation of structural disc changes, including disc height, signal intensity, and degenerative features, assessed at predefined follow-up intervals.

OTHER OUTCOMES:
Change From Baseline in EQ-5D-5L Index Score | From baseline to 24 months after the procedure
  Outcome Measure Description:
  EQ-5D-5L is a standardized measure of health-related quality of life across five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression). The index score is derived from the five-digit health state.

CONTACTS AND LOCATIONS:
Locations (1):
- Poliklinika Terasa, Košice, Košice Region, Slovakia